CLINICAL TRIAL: NCT01566422
Title: Comparative Effectiveness and Cost-Benefit Analysis of Vancomycin Powder in High Risk Spine Surgery Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: unable to enroll any participants
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Vanc-1510
Record Dates: First submitted 2012-03-12; First posted 2012-03-29 (Estimated); Last update posted 2018-04-20 (Actual); Status verified 2018-04

CONDITIONS: Surgical Site Infection
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vancomycin powder (Experimental): 80 randomized patients will be given vancomycin powder in the surgical sites prior to closure following spinal surgery.
  Interventions: Drug: Vancomycin powder
- Control (No Intervention): 80 participants who were not randomized to receive Vancomycin powder will receive no intervention at the conclusion of their surgery.

INTERVENTIONS:
Drug: Vancomycin powder — patients randomized to this group will receive vancomycin powder in the surgical incision after posterior spinal fusion.
  Arms: Vancomycin powder

SUMMARY:
Despite the use of prophylactic systemic antibiotics and improved surgical technique, surgical site infections remain a serious concern. The incidence of deep infection after spine surgery has been lowered with systemic antibiotics, yet after instrumented fusion for traumatic injuries infection rates remain as high as 10%. The impact on patients and cost of treating such infections is profound. With diminishing healthcare dollars and policy that refuses to reimburse for postoperative infections, it is critical that physicians and hospital systems seek out cost effective ways of decreasing postoperative infections. Local delivery of antibiotics into the surgical site have been found to significantly decrease infection rates in those undergoing posterior spine fusion for traumatic injuries as studied in a retrospective manner by the investigators of this grant. In this proposal the investigators will prospectively randomize patients undergoing posterior spinal stabilization for traumatic injuries into either receiving vancomycin powder into the surgical site (treatment) versus not receiving vancomycin powder (control) and subsequently follow infection rate, complications, and cost of care. The investigator's hypothesis is that i) vancomycin powder will decrease infection rates ii) have no systemic toxicity iii) and be a cost saving advancement in the safety of delivering spine surgical care.

ELIGIBILITY:
Inclusion Criteria

* All English-speaking patients ≥ 18 years undergoing posterior spine fusions at Vanderbilt University Medical Center for the treatment of traumatic injuries will be considered for inclusion

Exclusion Criteria

* have a known allergy to vancomycin
* do not agree to participate
* had previous spine surgery at the injury level within 6 months
* are pregnant
* have a history of Steven's Johnson Syndrome
* have a history of infections at the surgical site
* have a history of cancer or radiation treatment at the injured level
* have open spine fractures
* have traumatic injuries to non-spine organ systems that limit their functional capacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Determine efficacy of using local vancomycin powder | 2 years
  Patient demographics and perioperative information obtained will include: comorbidities known to increase the risk of infection, body mass index, level of injury, presence of neurologic deficit, prealbumin level, evidence of an open fracture elsewhere, injury severity score, operative time, estimated blood loss, and blood creatinine levels. All wounds will be assessed 4-6 weeks after surgery to address early surgical site infection (SSI).

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Background] Bibbo C, Patel DV. The effect of demineralized bone matrix-calcium sulfate with vancomycin on calcaneal fracture healing and infection rates: a prospective study. Foot Ankle Int. 2006 Jul;27(7):487-93. doi: 10.1177/107110070602700702. PMID 16842714
- [Background] Branstetter JG, Jackson SR, Haggard WO, Richelsoph KC, Wenke JC. Locally-administered antibiotics in wounds in a limb. J Bone Joint Surg Br. 2009 Aug;91(8):1106-9. doi: 10.1302/0301-620X.91B8.22216. PMID 19651846
- [Background] Buchholz HW, Engelbrecht H. [Depot effects of various antibiotics mixed with Palacos resins]. Chirurg. 1970 Nov;41(11):511-5. No abstract available. German. PMID 5487941
- [Background] Burdon DW. Principles of antimicrobial prophylaxis. World J Surg. 1982 May;6(3):262-7. doi: 10.1007/BF01653540. No abstract available. PMID 7113232
- [Background] Calderone RR, Garland DE, Capen DA, Oster H. Cost of medical care for postoperative spinal infections. Orthop Clin North Am. 1996 Jan;27(1):171-82. PMID 8539047
- [Background] Cavanaugh DL, Berry J, Yarboro SR, Dahners LE. Better prophylaxis against surgical site infection with local as well as systemic antibiotics. An in vivo study. J Bone Joint Surg Am. 2009 Aug;91(8):1907-12. doi: 10.2106/JBJS.G.01237. PMID 19651948
- [Background] Dahners LE, Funderburk CH. Gentamicin-loaded plaster of Paris as a treatment of experimental osteomyelitis in rabbits. Clin Orthop Relat Res. 1987 Jun;(219):278-82. PMID 3581579
- [Background] Edin ML, Miclau T, Lester GE, Lindsey RW, Dahners LE. Effect of cefazolin and vancomycin on osteoblasts in vitro. Clin Orthop Relat Res. 1996 Dec;(333):245-51. PMID 8981903
- [Background] Gitelis S, Brebach GT. The treatment of chronic osteomyelitis with a biodegradable antibiotic-impregnated implant. J Orthop Surg (Hong Kong). 2002 Jun;10(1):53-60. doi: 10.1177/230949900201000110. PMID 12401922
- [Background] Glassman SD, Dimar JR, Puno RM, Johnson JR. Salvage of instrumental lumbar fusions complicated by surgical wound infection. Spine (Phila Pa 1976). 1996 Sep 15;21(18):2163-9. doi: 10.1097/00007632-199609150-00021. PMID 8893444
- [Background] Gold HS, Moellering RC Jr. Antimicrobial-drug resistance. N Engl J Med. 1996 Nov 7;335(19):1445-53. doi: 10.1056/NEJM199611073351907. No abstract available. PMID 8875923
- [Background] O'Neill KR, Smith JG, Abtahi AM, Archer KR, Spengler DM, McGirt MJ, Devin CJ. Reduced surgical site infections in patients undergoing posterior spinal stabilization of traumatic injuries using vancomycin powder. Spine J. 2011 Jul;11(7):641-6. doi: 10.1016/j.spinee.2011.04.025. Epub 2011 May 19. PMID 21600853